CLINICAL TRIAL: NCT00846638
Title: Screening and Brief Intervention for Problem Drinking Women
Brief Title: Women's Health Habits Study
Acronym: WHHS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Grace Chang, MD, MPH, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIAAA-Chang-AA014678; R01AA014678 (NIH); NIH Grant R01AA014678
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Risk Drinking,Diabetes, Hypertension, Osteoporosis, Infertility
Keywords: Risk drinking; Women; Medical problems
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Osteoporosis; Infertility | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Diagnostic assessment with brief intervention and 3, 6, and 12 month follow-up
  Interventions: Behavioral: Brief Intervention
- 2 (Active Comparator): Diagnostic assessment with 12 month follow-up
  Interventions: Behavioral: Diagnostic assessment

INTERVENTIONS:
Behavioral: Brief Intervention — Diagnostic assessment followed by a single session Brief Intervention with 3, 6, and 12 month follow-up
  Arms: 1
Behavioral: Diagnostic assessment — Single session diagnostic assessment with 12 month followup
  Arms: 2

SUMMARY:
The purpose of this randomized trial is to test the effectiveness of screening and brief intervention for risk drinking by nonpregnant women with specific medical problems exacerbated by excessive alcohol consumption. The medical problems are female factor infertility, hypertension, diabetes, and osteoporosis, conditions that are costly to treat and difficult to manage. Just as pregnant women are thought to be highly motivated to modify their alcohol consumption, so women with specific medical problems worsened by alcohol intake are an appropriate group to receive a brief intervention.

ELIGIBILITY:
Inclusion Criteria:

- 1. has diabetes, hypertension, osteoporosis, or infertility 2. Not currently receiving treatment for alcohol or drug problems or substance related medical illness 3. Not currently experiencing physical dependence on alcohol, requiring medically supervised detoxification 4. Not currently abusing or physically dependent on opiates, cocaine, or other illicit drugs 5. Not currently pregnant. Subjects with infertility may become pregnant during the course of the study.

6. Not currently nursing. 7. Able to complete study measures.

Exclusion Criteria:

1. Alcohol screen negative or drinks within NIAAA sensible drinking limits for women
2. Does not agree to randomization and study terms

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2005-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Drinking outcome | 12 months post enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States